CLINICAL TRIAL: NCT00836498
Title: V260-027 Safety and Immunogenicity of RotaTeq™ in Elderly Subjects
Brief Title: A Study of the Safety and Immune Response to RotaTeq™ Vaccine in the Elderly (V260-027)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision not to pursue indication due to lack of demonstrable medical need
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-027; 2007_537
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Rotavirus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part I, RotaTeq (Experimental): 3 doses of RotaTeq
  Interventions: Biological: Comparator: RotaTeq
- Part I, placebo (Placebo Comparator): 3 doses of placebo
  Interventions: Biological: Comparator: Placebo
- Part II, RotaTeq (Experimental): 3 doses of RotaTeq
  Interventions: Biological: Comparator: RotaTeq
- Part II, RotaTeq and placebo (Experimental): 1 dose of RotaTeq and 2 doses of placebo
  Interventions: Biological: Comparator: RotaTeq + Placebo
- Part II, placebo (Placebo Comparator): 3 doses of placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Comparator: RotaTeq — Three 2.0 mL oral doses of RotaTeq. Vaccination 1 administered on Day 1, Vaccination 2 administered 28-42 days after Vaccination 1, and Vaccination 3 administered 28-42 days after Vaccination 2.
  Arms: Part I, RotaTeq; Part II, RotaTeq
Biological: Comparator: Placebo — Three 2.0 mL oral doses of RotaTeq. Vaccination 1 administered on Day 1, Vaccination 2 administered 28-42 days after Vaccination 1, and Vaccination 3 administered 28-42 days after Vaccination 2.
  Arms: Part I, placebo; Part II, placebo
Biological: Comparator: RotaTeq + Placebo — One 2.0 mL oral dose of RotaTeq and two 2.0 mL oral doses of placebo over an approximately 3-5 month treatment period
  Arms: Part II, RotaTeq and placebo

SUMMARY:
This is a Phase I clinical trial including 2 parts to evaluate the safety and immune response to RotaTeq™ /placebo in subjects of 65 to 80 years of age. In Part I, approximately 60 subjects in US will be randomly assigned to 1 of 2 treatment groups receiving 3 doses of RotaTeq™ or placebo. In Part II, approximately 200 subjects internationally will be randomly assigned to 1 of 3 treatment groups. Part II will start after Part I data analysis is reviewed and approved by the FDA/CBER, the Safety Evaluation Committee (SEC) and other regulatory agencies. Duration for the entire study will be approximately 4 years.

Note: As the result of a business decision by the Sponsor, the study did not proceed with Part II. Therefore, this report includes the results for Part I only.

ELIGIBILITY:
Inclusion Criteria:

* Is 65 to 80 years of age with controlled chronic illness
* agrees to participate in the study by giving written informed consent and cognitively competent as assessed by Mini-Mental State Examination
* for Part I: subject is living independently outside any long-term care facilities; for Part II: subject is expected to be a resident in a long term care facility (LTCF) including nursing homes with the exception of hospice care
* can be adequately followed for safety via visit or phone
* subject's routine safety lab results are within specified ranges
* has negative test results for HIV, Hepatitis B, and Hepatitis C

Exclusion Criteria:

* abdominal cancer/surgery within the past 6 months
* known or suspected immune diseases, e.g. diabetes
* any chronic or relapsing infections
* a fever at the time of immunization
* active vomiting or diarrhea at the time of immunization
* chronic diarrhea, irritable bowel syndrome, or inflammatory disease of intestinal or colon in the past 12 months
* subjects' spouses/cohabitants are not healthy or are immunocompromised; roommates in LTCFs are not healthy and/or do not agree to participate in the study
* cannot be adequately followed for safety via visit or phone
* any other clinically significant conditions that, in the investigators' opinion, would interfere with subject's participation in the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lawrence J, He S, Martin J, Schodel F, Ciarlet M, Murray AV. Safety and immunogenicity of pentavalent rotavirus vaccine in a randomized, double-blind, placebo-controlled study in healthy elderly subjects. Hum Vaccin Immunother. 2014;10(8):2247-54. doi: 10.4161/hv.29107. PMID 25424929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of participants occurred at 8 study sites in the United States.
Pre-assignment Details: Part II was not conducted; no participants were recruited.
Groups:
- RotaTeq™: Three dose regimen of RotaTeq™. Vaccination 1 administered on Day 1, Vaccination 2 administered 28-42 days after Vaccination 1, and Vaccination 3 administered 28-42 days after Vaccination 2.
- Placebo: Three dose regimen of matching placebo. Vaccination 1 administered on Day 1, Vaccination 2 administered 28-42 days after Vaccination 1, and Vaccination 3 administered 28-42 days after Vaccination 2.
Period: Overall Study
Arm/Group | RotaTeq™ | Placebo
Started | 44 | 22
Completed | 40 (Participant who discontinued the study vaccination due to AE completed the 180-day safety follow-up.) | 21
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ | Placebo | Total
Number analyzed (Participants) | 44 | 22 | 66
Age, Customized [Number; unit: participants] — Between 65 and 80 years.
  participants | 44 | 22 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 21 | 9 | 30
Region of Enrollment [Number; unit: participants]
  United States | 44 | 22 | 66

OUTCOME MEASURES:

1. Primary Outcome: Part I: Number of Participants With Nonserious and Serious Adverse Experiences (AEs)
Description: All randomized participants were contacted via telephone or in-center visit on Days 7, 14, 28, and 42 after each dose. Participants received a Vaccination Report Card (VRC) at each vaccination visit as well as instructions for recording AEs. Participants were also instructed to record potential acute gastroenteritis episodes (AGEs) that occurred within 42 days after any dose on the report card.
Time Frame: Up to 42 days following any dose of RotaTeq™ or placebo
Population: All randomized participants who received at least one dose of RotaTeq™ or placebo are included in the summaries.
  Number of participants with one or more adverse experience.
Measure: Number; unit: participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 44 | 22
participants | 26 | 9

2. Primary Outcome: Part I: Number of Participants With Serious Adverse Experiences (SAEs)
Description: All randomized participants were contacted via telephone or in-center visit on Days 7, 14, 28, and 42 after each dose. Participants received a Vaccination Report Card (VRC) at each vaccination visit as well as instructions for recording AEs. Participants were also instructed to record potential acute gastroenteritis episodes (AGEs) that occurred within 42 days after any dose on the report card.
  SAEs were followed by passive surveillance (in which either participants self reported or information was collected at participants' last visit) for 180 days following the final dose.
Time Frame: Up to 180 days following the third dose of RotaTeq™ or placebo
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 40 | 21
participants | 1 | 0

3. Primary Outcome: Part I: Geometric Mean Titers (GMT) of Serum Anti-rotavirus Immunoglobulin A (IgA)
Description: GMTs of serum anti-rotavirus IgA responses after 1, 2, or 3 doses of RotaTeq™ or placebo.
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: All endpoints exclude protocol violators & participants with invalid data based on laboratory determinations.
  Analyses of endpoints based on a Per-protocol (PP) population: participants who received at least one dose study designed material and had at least one valid assay result within study specified time window & were not protocol violators.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n=36 RotaTeq/ n=19 placebo) | 679.6 [464.5 to 994.2] | 578.4 [361.1 to 926.4]
  Postdose 1 GMT (n=28 RotaTeq/ n=16 placebo) | 1026.8 [621.6 to 1696.2] | 552.8 [314.5 to 971.8]
  Postdose 2 GMT (n=37 RotaTeq/ n=20 placebo) | 1187.0 [807.6 to 1744.5] | 657.7 [404.9 to 1068.5]
  Postdose 3 GMT (n=38 RotaTeq/ n=18 placebo) | 1179.9 [785.5 to 1772.2] | 578.5 [349.0 to 959.0]

4. Primary Outcome: Part II: Number of Participants With Nonserious Adverse Experiences
Description: Part II was not conducted due to study termination; this report summarizes study results from Part I only.
Time Frame: Up to 42 days following any dose of RotaTeq™ and/or placebo
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Part II: Number of Participants With Serious Adverse Experiences
Description: Part II was not conducted due to study termination; this report summarizes study results from Part I only.
Time Frame: Up to 180 days following the third dose of RotaTeq™ and/or placebo
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part I: Geometric Mean Titer (GMT) of Serum Neutralizing Antibody (SNA) Response to Human Rotavirus Serotype G1
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- RotaTeq: Three dose regimen of RotaTeq™. Vaccination 1 administered on Day 1, Vaccination 2 administered 28-42 days after Vaccination 1, and Vaccination 3 administered 28-42 days after Vaccination 2.
Arm/Group | RotaTeq | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n=36 RotaTeq/ n=19 Placebo) | 314.5 [219.2 to 451.3] | 281.4 [152.6 to 519.1]
  Postdose 1 GMT (n=28 RotaTeq/ n=16 Placebo) | 506.2 [330.5 to 775.4] | 228.7 [121.0 to 432.4]
  Postdose 2 GMT (n=37 RotaTeq/ n=20 Placebo) | 556.1 [389.8 to 793.5] | 226.7 [136.8 to 375.6]
  Postdose 3 GMT (n=38 RotaTeq/ n=18 Placebo) | 535.9 [395.9 to 725.4] | 231.6 [140.3 to 382.3]

7. Secondary Outcome: Part I: Geometric Mean Titer (GMT) of Serum Neutralizing Antibody (SNA) Response to Human Rotavirus Serotype G2
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RotaTeq | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n= 36 RotaTeq/ n=19 placebo) | 62.8 [43.6 to 90.5] | 68.2 [40.6 to 114.6]
  Postdose 1 GMT (n= 28 RotaTeq/ n=16 placebo) | 123.4 [81.4 to 187.2] | 56.3 [34.5 to 92.0]
  Postdose 2 GMT (n= 37 RotaTeq/ n=20 placebo) | 111.2 [81.6 to 151.6] | 74.3 [46.2 to 119.5]
  Postdose 3 GMT (n= 38 RotaTeq/ n=18 placebo) | 127.0 [93.1 to 173.3] | 71.3 [44.5 to 114.3]

8. Primary Outcome: Part II: Geometric Mean Titer (GMT) of Serum Anti-rotavirus Immunoglobulin A (IgA)
Description: Part II was not conducted due to study termination; this report summarizes study results from Part I only.
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Part I: Geometric Mean Titer (GMT) of Serum Neutralizing Antibody (SNA) Response to Human Rotavirus Serotype G3
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RotaTeq | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n= 36 RotaTeq/ n=19 placebo) | 141.8 [95.7 to 210.1] | 90.9 [62.1 to 133.0]
  Postdose 1 GMT (n= 28 RotaTeq/ n=16 placebo) | 404.6 [230.6 to 710.0] | 94.5 [59.4 to 150.4]
  Postdose 2 GMT (n= 37 RotaTeq/ n=20 placebo) | 330.7 [219.5 to 498.3] | 119.8 [79.6 to 180.2]
  Postdose 3 GMT (n= 38 RotaTeq/ n=18 placebo) | 388.0 [264.7 to 568.7] | 102.1 [66.3 to 157.3]

10. Secondary Outcome: Part I: Geometric Mean Titer (GMT) of Serum Neutralizing Antibody (SNA) Response to Human Rotavirus Serotype G4
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RotaTeq | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n= 36 RotaTeq/ n=19 placebo) | 91.6 [66.1 to 126.8] | 102.7 [65.7 to 160.4]
  Postdose 1 GMT (n= 28 RotaTeq/ n=16 placebo) | 199.2 [128.5 to 308.6] | 93.1 [55.4 to 156.2]
  Postdose 2 GMT (n= 37 RotaTeq/ n=20 placebo) | 223.9 [154.2 to 325.3] | 110.1 [68.4 to 177.5]
  Postdose 3 GMT (n= 3 RotaTeq/ n=18 placebo) | 221.7 [162.9 to 301.7] | 106.9 [64.2 to 178.0]

11. Secondary Outcome: Part I: Geometric Mean Titer (GMT) of Serum Neutralizing Antibody (SNA) Response to Human Rotavirus Serotype P1A[8]
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3 of RotaTeq™ or placebo
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RotaTeq | Placebo
Number analyzed (Participants) | 44 | 22
titers
  Pre-Vaccination GMT (n= 36 RotaTeq/ n=19 placebo) | 230.8 [166.8 to 319.4] | 143.4 [88.9 to 231.3]
  Postdose 1 GMT (n= 28 RotaTeq/ n=16 placebo) | 306.4 [219.8 to 427.0] | 126.1 [78.7 to 202.0]
  Postdose 2 GMT (n= 37 RotaTeq/ n=20 placebo) | 375.6 [278.4 to 506.6] | 154.0 [98.0 to 241.9]
  Postdose 3 GMT (n= 38 RotaTeq/ n=18 placebo) | 327.6 [253.8 to 423.0] | 160.7 [102.3 to 252.3]

12. Secondary Outcome: Part II: Geometric Mean Titers (GMTs) of Serum Neutralizing Antibody (SNA) Responses to G1, G2, G3, G4, and P1A
Description: Part II was not conducted due to study termination; this report summarizes study results from Part I only.
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part II: Percentage of Participants With a >=3-fold Rise From Baseline of Serum Anti-rotavirus IgA and SNA Responses to Rotavirus Serotypes G1, G2, G3, G4 and P1A
Description: Part II was not conducted due to study termination; this report summarizes study results from Part I only.
Time Frame: Prior to Dose 1 and 28 to 42 days Postdose 1, 2, and 3
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | RotaTeq™ | Placebo
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/22
Other Adverse Events (participants affected / at risk) | 18/44 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ (N=44) | Placebo (N=22)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) — Reported within the 43-180 days post vaccination 3
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) — Reported within the 42-day period post vaccination 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ (N=44) | Placebo (N=22)
Diarrhoea (Gastrointestinal disorders) | 11 (16) | 2 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (10) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (3)
Headache (Nervous system disorders) | 7 (14) | 4 (9)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less